CLINICAL TRIAL: NCT00510354
Title: Multicenter, Single-arm, Two Stage Phase II Trial of RAD001 (Everolimus) With Imatinib in Imatinib-resistant Patients With Progressive GIST
Brief Title: Treatment of Patients With Everolimus and Imatinib Mesylate Who Have Progressive Gastro Intestinal Stromal Tumors (GIST) and Are Resistant to Imatinib Mesylate
Acronym: Radix
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001C2454; 2005-004837-16
Record Dates: First submitted 2007-07-31; First posted 2007-08-02 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2016-11

CONDITIONS: Progressive Gastrointestinal Stromal Tumor
Keywords: Progressive GIST; Resistance to Imatinib mesylate
MeSH Terms: interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RAD001 + Imatinib (Experimental)
  Interventions: Drug: Imatinib mesylate

INTERVENTIONS:
Drug: Imatinib mesylate

SUMMARY:
The purpose of this multicenter, single-arm, Simon two-stage, phase II trial is to determine the efficacy and safety of everolimus in combination with Imatinib mesylate in patients with previously treated, histologically proven GIST whose disease has recurred or progressed while receiving 400 mg/day of Imatinib mesylate at any time during at least a 2 months' treatment period.

ELIGIBILITY:
Inclusion criteria:

1. Histological proven diagnosis of GIST
2. Objectively documented evidence of progressive disease according to the RECIST criteria despite at least 2 months' continuous treatment with Imatinib mesylate at a dosage of 400 mg/day
3. Clinical evidence of resistance to Imatinib mesylate on treatment with 400 mg/day Imatinib
4. Progression must be documented on CT or MRI scans. The scans on which progression is documented should be at maximum 2 weeks old. New scans are only required as baseline scans if they are older then approx. 2 weeks
5. At least one measurable lesion (longest diameter ≥ 20 mm on conventional CT or MRI scan; ≥ 10 mm on spiral CT)
6. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
7. Adequate bone marrow, liver and renal function on Imatinib treatment
8. Patients must be at least 4 weeks since prior major surgery and recovered, at least 2 weeks since prior minor surgery and recovered

Exclusion criteria:

1. Female patients who are pregnant or breast feeding, or patients of reproductive potential not employing an effective method of birth control. Because oral, implantable or injectable contraceptives may be affected by cytochrome P450 interactions, an appropriate method of birth control should be used throughout the trial in both sexes. Women of childbearing potential must have a negative serum pregnancy test ≤ 48 hours prior to the administration of study medication
2. Patients presenting with known or symptomatic CNS metastases or leptomeningeal involvement
3. Use of other investigational cancer therapies within 28 days prior to enrollment or which are currently being or planned to be received during the course of the study
4. Patients who previously received rapamycin in combination with Imatinib
5. Patients with any concurrent major medical condition liable to compromise the patient's participation in the study (e.g. known HIV infection, uncontrolled diabetes, serious cardiac dysrhythmia or condition, New York Heart Association classification of III or IV, congestive cardiac failure, myocardial infarction within 6 months, unstable angina, chronic or acute renal or liver disease, uncontrolled infections including abscess or fistulae, etc.)
6. Patients with a history of another malignancy within 5 years prior to study entry, except curatively treated non-melanotic skin cancer or in-situ cervical cancer
7. Patients receiving glucocorticoids (only if the p70s6 kinase-1 assay is being performed), since glucocorticoids have been shown to inhibit p70s6 kinase-1 activity

Other protocol defined inclusion/ exclusion criteria may apply

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Tumor assessments should be performed by a CT or MRI scan after 4 months. Response to treatment with RAD001 plus Imatinib mesylate at 4 months (defined as progression-free survival (PFS) at 4 months). | at 4 months

SECONDARY OUTCOMES:
Tolerability and safety assessed by AEs and SAEs. Objective tumor response rate (complete response [CR] and partial response [PR]) assessed by CT or MRI PFS at month 12 for patients with data available from follow up observation (optional) | At 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Germany (7):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Frankfurt/M
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Tübingen